CLINICAL TRIAL: NCT00836277
Title: Phase II Study of Irinotecan and Panitumumab as Second-Line Therapy for Patients With Advanced Esophageal Adenocarcinoma
Brief Title: Phase II Study of Irinotecan and Panitumumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weijing Sun, MD, FACP (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Weijing Sun, MD, FACP, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-161
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-09

CONDITIONS: Esophageal Cancer
Keywords: Panitumumab; Irinotecan; Esophageal Adenocarcinoma; Phase II
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Panitumumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan plus panitumumab (Experimental): Irinotecan 100 mg/m2 IV Day 1 and Day 8
  + Panitumumab 9mg/kg IV Day 1 Cycle = 21 days
  Interventions: Drug: Panitumumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Panitumumab — 9mg/kg IV Day 1 Cycle = 21 days
  Other Names: ABX-EGF
Drug: Irinotecan — 125mg/m2 IV Day 1 and Day 8
  Other Names: Camptosar; Campto; CPT-11

SUMMARY:
This study proposes a single-arm, phase II study of irinotecan with panitumumab as second-line therapy for patients with advanced esophageal adenocarcinoma. Efficacy will be assessed by response rate, with an exploratory outcome endpoint of time to progression (as panitumumab may result in prolonged stable disease). In addition to the usual safety assessments, molecular correlates will be carried out in order to search for pharmacodynamic and pharmacogenomic features that may correlate with response. Measures of host/patient immune function will be assessed by evaluating the relationship between Fc receptor polymorphisms and response in patients treated with panitumumab. Measures of EGFR protein and phosphoprotein expression by immunohistochemical- (IHC-) staining, K-ras mutation status1 and reverse-phase protein arrays (RPPA) and EGFR gene amplification by fluorescence in situ hybridization (FISH) will be assessed as exploratory correlates.

DETAILED DESCRIPTION:
Esophageal cancer is a highly lethal malignancy that is increasing in incidence, especially the histologic subtype of adenocarcinoma. Fully 50% of patients present with advanced, incurable disease. Of the remainder who are diagnosed at curable stages, at most 30% are long-term survivors. Advances in therapy for both local and advanced disease have been stagnant in the past few decades. As such, there is an urgent need for advances in therapy. The development of modern cytotoxic chemotherapy and in particular, biologically targeted agents, provides hope for improving the outcome in these patients.

The semi-synthetic derivative of camptothecin, irinotecan, is active in esophageal adenocarcinoma, both alone and in combination with cisplatin. Use as front-line therapy in both multi-modality regimens and combination chemotherapy is common. More recently, the elucidation of the role of the epidermal growth factor receptor (EGFR) pathway in esophageal cancer has resulted in the pre-clinical and clinical study of the activity of EGFR directed agents for treatment of esophageal cancer.

The anti-EGFR antibodies, panitumumab and cetuximab, are active as both single agents and in combination with cytotoxic chemotherapy in patients with colorectal adenocarcinoma. In particular, the combination of irinotecan and cetuximab is active for irinotecan refractory colorectal cancer, while panitumumab is active compared with best supportive care. In our clinic, we have empiric evidence for the unexpectedly significant activity of the combination of cetuximab and irinotecan as third-line treatment for advanced esophageal adenocarcinoma. Panitumumab has the clinical advantages, compared with cetuximab, of being fully human,, thus resulting in a lower frequency of infusion reactions.

This recent experience with these targeted agents in solid tumors, while still promising, has yielded relatively modest results.7-11 Notably, however, retrospective analyses of clinical trials are consistently revealing that differences in treatment effect between subgroups of patients can be associated with specific molecular profiles.12-18 These findings suggest the potential for a more rational approach to trial design that would use patient and tumor characteristics to select patients for therapy, thus enriching the population of responders.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of locally recurrent or metastatic adenocarcinoma of the esophagus which is incurable with standard therapy.
* Patients must have measurable disease outside a previous radiation port, or which has developed in the port since the conclusion of radiation and is biopsy-proven to be recurrent cancer.
* One prior chemotherapy regimen for metastatic disease, with the exception of prior irinotecan or panitumumab.
* Prior radiation therapy to no more than 20% of the bone marrow is allowed. No treatment with wide field radiation within 4 weeks of entry onto this study.
* Full recovery from the effects of any prior surgery.
* Man or woman >18 years of age.
* ECOG performance status <2 (Karnofsky >60%)
* Life expectancy of >3 months
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Hemoglobin ≥ 9.0 g/dL
* Creatinine < or = to 1.5 mg/dL
* Creatinine clearance > or = to 50 mL/min calculated by the Cockcroft-Gault method as follows:
* Male creatinine clearance = (140 - age) x (weight in Kg) / (serum Cr x 72)
* Female creatinine clearance = (140 - age) x (weight in Kg) x 0.85 / (serum Cr x 72)
* Aspartate aminotransferase (AST) < or = to 3 x ULN (if liver metastases less than or equal to 5 x ULN)
* Alanine aminotransferase (ALT) < or = to 3 x ULN (if liver metastases less than or equal to 5 x ULN)
* Total bilirubin < or = to 1.5 x ULN
* Magnesium ≥ lower limit of normal
* Potassium > or = to lower limit of normal
* Because the effects of irinotecan and panitumumab on the developing human fetus are unknown, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* History or known presence of central nervous system (CNS) metastases unless CNS metastases have been irradiated and are stable.
* History of another primary cancer, except:
* Curatively treated in situ cervical cancer
* Curatively resected non-melanoma skin cancer
* Other primary solid tumor curatively treated with no known active disease present and no treatment administered for greater than or equal to 5 years prior to enrollment
* Pre-existing peripheral neuropathy > grade 1.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to panitumumab or irinotecan.
* Patients receiving any medications or substances that are established or probable inhibitors or inducers of P450 3A4 are ineligible.
* Prior anti-EGFr antibody therapy (eg, cetuximab) or treatment with small molecule EGFr inhibitors (eg, gefitinib, erlotinib, lapatinib)
* Radiotherapy < or = to 14 days prior to enrollment.
* Systemic chemotherapy, hormonal therapy, immunotherapy, or experimental or approved proteins/antibodies (or small molecules for Phase I studies) (eg, bevacizumab)< or = to 30 days before enrollment
* Subjects requiring chronic use of immunosuppressive agents (eg, methotrexate, cyclosporine)
* Any investigational agent or therapy < or = to 30 days before enrollment
* Prior therapy with Irinotecan or panitumumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of interstitial lung disease (e.g. pneumonitis or pulmonary fibrosis) or any evidence of interstitial lung disease on baseline chest CT scan
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.
* Women who test positive for serum or urine pregnancy test < 72 hours before randomization or is breast feeding
* Known positive test(s) for acute or chronic active hepatitis B infection
* Major surgery within 28 days or minor surgery within 14 days of study enrollment
* Men or women of child-bearing potential (women who are post-menopausal < 52 weeks, not surgically sterilized, or not abstinent) not consenting to use adequate contraception (per institutional standard of care) during treatment and for six months after the last investigational product(s) administration
* Any underlying condition which in the opinion of the principal investigator will interfere with safety or with compliance with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weijing Sun, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Yoon H, Karapetyan L, Choudhary A, Kosozi R, Bali GS, Zaidi AH, Atasoy A, Forastiere AA, Gibson MK. Phase II Study of Irinotecan Plus Panitumumab as Second-Line Therapy for Patients with Advanced Esophageal Adenocarcinoma. Oncologist. 2018 Sep;23(9):1004-e102. doi: 10.1634/theoncologist.2017-0657. Epub 2018 May 16. PMID 29769385

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan + Panitumumab: Participants with a diagnosis of locally recurrent and/or metastatic esophageal adenocarcinoma treated with panitumumab 9 mg/kg on day 1 and irinotecan 100 mg/m^2 on days 1 and 8 of each 21 day cycle to a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Irinotecan + Panitumumab
Started | 24
Completed | 18
Not Completed | 6
Not completed — Not evaluable for response | 6

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan + Panitumumab
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 62.5 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Response rate (RR) = the # participants with partial response (PR) + # participants with (CR) / # participants with (PR) + # participants with (CR ) + # participants with (SD) + # participants with (PD). This proportion was subsequently multiplied by 100. RECIST v1.0 criteria for Target Lesions was used: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Up to 14 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Irinotecan + Panitumumab
Number analyzed (Participants) | 18
percentage of participants | 6 [1 to 26]

2. Primary Outcome: Clinical Benefit Rate (CBR)
Description: Using RECIST v1.0 criteria, clinical benefit rate (CBR) = # participants with (PR) + # participants with (CR) + # participants with (SD) / # participants with (PR) + # participants with (CR) + # participants with (SD) + # participants with (PD). This proportion was subsequently multiplied by 100. RECIST v1.0 criteria for Target Lesions is defined as: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 14 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Irinotecan + Panitumumab
Number analyzed (Participants) | 18
percentage of participants | 50 [29 to 71]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Survival time the is free of disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 45 months (cohort)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan + Panitumumab
Number analyzed (Participants) | 18
months | 2.9 [1.6 to 5.3]

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 45 months (cohort)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan + Panitumumab
Number analyzed (Participants) | 18
months | 7.2 [4.1 to 8.9]

5. Secondary Outcome: 1-year (Overall) Survival Rate
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Irinotecan + Panitumumab
Number analyzed (Participants) | 18
percentage of participants | 11.1

ADVERSE EVENTS:
Arm/Group | Irinotecan + Panitumumab
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan + Panitumumab (N=18)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Weight loss (General disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Perforation, GI, Small bowel NOS (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Infection with unknown ANC, Catheter-related (Infections and infestations) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan + Panitumumab (N=18)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 5
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 10
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 13
Hemoglobin (Blood and lymphatic system disorders) | 15
Cardiac General - Other (Specify, __) (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 3
Hypotension (Cardiac disorders) | 4
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1
Insomnia (General disorders) | 3
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 1
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 12
Dehydration (Gastrointestinal disorders) | 1
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Stricture/stenosis (including anastomotic), GI, Esophagus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 5
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 9
Hemorrhage, pulmonary/upper respiratory, Nose (Blood and lymphatic system disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Infection with unknown ANC, Catheter-related (Infections and infestations) | 1
Infection with unknown ANC, Mucosa (Infections and infestations) | 1
Edema: limb (Blood and lymphatic system disorders) | 2
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6
Alkaline phosphatase (Metabolism and nutrition disorders) | 7
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 9
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 11
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13
Muscle weakness, generalized or specific area (not due to neuropathy), Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Mood alteration, Anxiety (Nervous system disorders) | 3
Mood alteration, Depression (Nervous system disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 5
Eyelid dysfunction (Eye disorders) | 1
Pain, Esophagus (General disorders) | 1
Pain, Extremity-limb (General disorders) | 1
Pain, Head/headache (General disorders) | 1
Pain, Oral-gums (General disorders) | 1
Pain, Throat/pharynx/larynx (General disorders) | 1
Pain, Tumor pain (General disorders) | 1
Pain, Bone (General disorders) | 2
Pain, Abdomen NOS (General disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes